CLINICAL TRIAL: NCT05013619
Title: Pain Prevalence, Distribution, Effect on Activities of Daily Life in Patients With Adolescent Cerebral Palsy and a Comparion of the Mother-child Report
Brief Title: Pain Prevalence, Distribution, Effect on Activities of Daily Life in Patients With Adolescent Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 20
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; adolescent; pain; parent report; self report
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescent cerebral palsy: Demographical data, the subtypes of CP, Gross Motor Functional Classification System level, circumstances of pain, pain questionnaire will be analyzed.
  Interventions: Other: Circumstances of pain; Other: Pain Questionnaire; Other: Gross Motor Functional Classification System; Other: The subtypes of Cerebral palsy
- adolescent cerebral palsy's mother: pain questionnaire will be analyzed.
  Interventions: Other: Pain Questionnaire

INTERVENTIONS:
Other: Circumstances of pain — It will be questioned in which situations the pain occurred in the previous week (at rest from spasms, at rest from splints, on feeding, on moving, on dressing, at night, on exercise, on other treatments, on botulinum toxin application) and record as yes/no.
  Groups: adolescent cerebral palsy
Other: Pain Questionnaire — Participants will be asked to respond to the initial question "Over the past month, have you experienced physical pain?" (yes or no). Those responding "yes" will be asked "Please indicate how severe your pain was over the past month, on average," with response options from 1 (very little pain) to 10 (extremely painful). They will be also asked to indicate "How much the pain gets in the way of your daily activities over the past month" from a low of 1 (does not get in the way at all) to 10 (unable to carry out activities because of the pain). Finally, they will be asked to indicate the body regions in which they experienced pain.
Other: Gross Motor Functional Classification System — Severity of CP will be determined based on the Gross Motor Functional Classification System (GMFCS). GMFCS is a standardised measure that classifies gross motor functions in children with CP. Children in level I are very independent in motor functions while those in level V are the least independent
  Groups: adolescent cerebral palsy
Other: The subtypes of Cerebral palsy — The subtypes of CP will be classified, using the Swedish classification, into spastic (tetraplegia, diplegia and hemiplegia), ataxic, dyskinetic and mixed
  Groups: adolescent cerebral palsy

SUMMARY:
Pain is the most common secondary condition in patients with CP and the most important factor associated with reduced health-related quality of life. Pain in adolescents with CP is reported approximately 50-75%. Despite being a condition that can be seen with such a high prevalence, it is difficult for researchers and clinicians to capture this subjective perception in CP, as the individual may be a small child, may be cognitively impaired, visually impaired, or have communication difficulties. For these reasons, unrecognized pain can have negative effects on quality of life and participation in daily living activities, both as a result of limited mobility resulting from pain itself and fear-driven avoidance of specific activities. Self-report of pain is appropriate for individuals with CP without cognitive impairment. However, depending on the severity of communication impairment, self-report may be limited or even impossible to obtain in individuals with severe CP. In the case of individuals with CP, self-report supplemented with parent report, when possible, is the recommended strategy.

The aims of this study: (i) to explore what is known about the prevalence, location, intensity and the effect of pain on daily lives of adolescents with CP; (ii) to demonstrate the relation between pain, clinical and sociodemographic characteristics; (iii) to compare self-reports of pain with mothers'reports of their child's pain.

DETAILED DESCRIPTION:
The investigators will record demographical data including age, gender, height (cm), weight (kg), body mass index (BMI), school type, type of family (core or combined family) of the children and socioeconomic status of the family, mothers' age and educational level. The subtypes of CP will be classified, using the Swedish classification, into spastic (tetraplegia, diplegia and hemiplegia), ataxic, dyskinetic and mixed. Severity of CP will be determined based on the Gross Motor Functional Classification System. It will be questioned in which situations the pain occurred in the previous week (at rest from spasms, at rest from splints, on feeding, on moving, on dressing, at night, on exercise, on other treatments, on botulinum toxin application) and record as yes/no. The pain questionnaire described by Doralp et al (14) will be used both for the self-evaluation of adolescents with CP' pain and for mothers to evaluate their children's pain. Participants will be asked to respond to the initial question "Over the past month, have you experienced physical pain?" (yes or no). Those responding "yes" will be asked "Please indicate how severe your pain was over the past month, on average," with response options from 1 (very little pain) to 10 (extremely painful). They will be asked to indicate "How much the pain gets in the way of your daily activities over the past month" from a low of 1 (does not get in the way at all) to 10 (unable to carry out activities because of the pain). Finally, they will be asked to indicate the body regions in which they experienced pain.

ELIGIBILITY:
Inclusion Criteria for patients:

* adolescents, aged 8 to 18 years with a diagnosis of cerebral palsy
* able to understand and answer the questions

Exclusion Criteria for patients:

* previous interventional procedures, such as surgery within the last one month
* using painkillers
* having concomittan diagnosed 'Autism Spectrum Disorder' or 'Attention Deficit Hyperactivity Disorder' or another neuromuscular disorder

Inclusion Criteria for their mothers:

* primary caregivers who spend most of their time with their children
* do not work outside the home

Exclusion Criteria for their mothers:

* not primary caregivers who spend most of their time with their children
* work outside the home

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescent cerebraly palsy and their mothers
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Functional Classification System level | Through study completion, an average of 1 month
  GMFCS is a standardised measure that classifies gross motor functions in children with CP. Children in level I are very independent in motor functions while those in level V are the least independent .
Pain distribution | Through study completion, an average of 1 month
  It will be questioned in which situations the pain occurred in the previous week (at rest from spasms, at rest from splints, on feeding, on moving, on dressing, at night, on exercise, on other treatments, on botulinum toxin application)
The pain questionnaire | Through study completion, an average of 1 month
  Participants will be asked to respond to the initial question "Over the past month, have you experienced physical pain?" (yes or no). Those responding "yes" will be asked "Please indicate how severe your pain was over the past month, on average," with response options from 1 (very little pain) to 10 (extremely painful). They will be also asked to indicate "How much the pain gets in the way of your daily activities over the past month" from a low of 1 (does not get in the way at all) to 10 (unable to carry out activities because of the pain). Finally, they will be asked to indicate the body regions in which they experienced pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özcan, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No